CLINICAL TRIAL: NCT06725381
Title: A Phase 1 Clinical Study of the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of SKB571 for Injection in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study of SKB571 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB571-I-01
Record Dates: First submitted 2024-11-28; First posted 2024-12-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Solid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental)
  Interventions: Drug: SKB571

INTERVENTIONS:
Drug: SKB571 — SKB571 for injection is administered every 3 weeks (q3w) until radiographic disease progression (PD), intolerable toxicity, death, or discontinuation of treatment, whichever occurs first.

SUMMARY:
This is a first-in-human (FIH), phase 1, multicenter, open-label study of SKB571 to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity in adult subjects with advanced or metastatic solid tumor .

DETAILED DESCRIPTION:
This is a first-in-human (FIH), phase 1, multicenter, open-label study of SKB571 to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity in adult subjects with advanced or metastatic solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-75 years at the time of signing the informed consent form
2. Subjects with histologically or cytologically confirmed locally advanced or metastatic solid tumors .
3. Subjects with at least one measurable lesion assessed by the investigator according to RECIST v1.1.
4. Subjects with Eastern Cooperative Oncology Group (ECOG) status score of 0 or 1.
5. Subjects who are assessed by the investigator to have an expected survival of ≥ 3 months.
6. Subjects who have adequate organ function.
7. Subjects who have recovered from all toxicities due to prior therapy .
8. Male and female subjects must agree to use highly effective contraception methods during the study treatment.
9. Subjects who voluntarily sign the informed consent form.

Exclusion Criteria:

1. Subjects with known active or untreated central nervous system (CNS) metastases.
2. Subjects with other malignant tumors within 3 years prior to the first dose.
3. Subjects with history of major cardiovascular, cerebrovascular, or thromboembolic disease.
4. Subjects with known active pulmonary tuberculosis.
5. Subjects with human immunodeficiency virus (HIV) infection, or any known active viral hepatitis, or hepatitis B or hepatitis C.
6. Subjects with major surgery within 28 days prior to the first dose.
7. Subjects with known allergy or hypersensitivity to SKB571 or its excipients.
8. Subjects with clinically severe lung injuries due to pulmonary complications.
9. Subjects with a history of allogeneic tissue/solid organ transplant.
10. Uncontrolled pleural effusion, pericardial effusion, or ascites effusion requiring repeated drainage.
11. Subjects who have received live vaccines within 30 days prior to the first dose of study treatment, or who are scheduled to receive live vaccines during the study.
12. Subjects who have received strong cytochrome P450 (CYP3A4) inhibitors or inducers, or BCRP inhibitors within 2 weeks prior to the first dose of study treatment or within 5 half-lives of known drug, whichever is longer.
13. Subjects who have received chemotherapy, immunotherapy, or biological therapy within 4 weeks prior to the first dose of study treatment.
14. Subjects with active infection requiring systemic anti-infective therapy within 14 days prior to the first dose of study treatment.
15. Subjects with any disease requiring systemic treatment with corticosteroids (prednisone at doses > 10 mg/d or similar drugs with equivalent doses) or other immunosuppressive therapy within 14 days prior to the first dose of study treatment.
16. Subjects have received an investigational agent or has used an investigational device within 28 days prior to initial dose administration of SKB571.
17. Subjects whose condition deteriorates rapidly before the first dose, such as a severe physical impariment or a change in ECOG score no longer meeting the inclusion criteria.
18. Subjects with a known history of psychosis or drug abuse that will preclude the subject from completing the study.
19. Any condition that, in the opinion of the investigator, will interfere with the assessment of study treatment or the safety of the subject or the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects achieving Dose-limiting toxicity (DLT) | From data of initial dose until up to 21 days for treatment
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  The sum of the number of cases with Complete Response (CR) and Partial Response (PR) in all treated tumor patients (CR + PR) divided by the total number of cases.
Progression Free Survival (PFS) | Up to 24 months
  Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
Duration of Response (DOR) | Up to 24 months
  Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
Overall Survival (OS) | Up to 24 months
  Time from start of treatment to death due to any reason.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Guangxi Medical University Cancer Hospital, Linyi, Shandong
  - Si Chuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Bei Jing Cancer Hospital, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Shanghai East Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Zhongshan Hospital, Shanghai